CLINICAL TRIAL: NCT00398671
Title: PreCoCa - "Prehospital Cooling With Cool-Caps"
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: PreCoCa-1
Record Dates: First submitted 2006-11-13; First posted 2006-11-14 (Estimated); Last update posted 2015-02-27 (Estimated); Status verified 2008-12

CONDITIONS: Heart Arrest
Keywords: primary successful cardio-pulmonary resuscitation; pre-hospital setting
MeSH Terms: conditions — Heart Arrest

INTERVENTIONS:
Device: Application of cool cap after primary successful CPR

SUMMARY:
This study shall investigate the feasibility of the use of cool-caps in the preclinical setting in patients with successful primary cardio-pulmonary resuscitation Hypothesis: cool-caps are efficient and feasible to use in the preclinical setting in patients after successful CPR.

ELIGIBILITY:
Inclusion Criteria:

* All patients with primary successful CPR

Exclusion Criteria:

* Age < 18
* Pregnancy
* Severe bleeding or severe trauma
* Body core temperature < 34 degrees celsius

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2006-01; Primary Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
Body core temperature at hospital/ ICU admission | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Dietrich Hasper, MD, Principal Investigator — Charite University Medicine
Locations (1):
- Charite University Hospital, Berlin, State of Berlin, Germany

REFERENCES:
- [Derived] Storm C, Schefold JC, Kerner T, Schmidbauer W, Gloza J, Krueger A, Jorres A, Hasper D. Prehospital cooling with hypothermia caps (PreCoCa): a feasibility study. Clin Res Cardiol. 2008 Oct;97(10):768-72. doi: 10.1007/s00392-008-0678-1. Epub 2008 May 29. PMID 18512093